CLINICAL TRIAL: NCT00005098
Title: Study of Genotype and Phenotype in Patients With Alpha 1-Antitrypsin Deficiency
Status: Terminated | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pittsburgh (Other)
Other Study IDs: 199/14810; WUSM-930603
Record Dates: First submitted 2000-04-06; First posted 2000-04-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-05

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: alpha 1-antitrypsin deficiency; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Genetic Diseases, Inborn; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Establish cell lines from patients with alpha 1-antitrypsin deficiency in order to examine genetic traits that predispose to liver injury.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo blood draw and skin biopsy. Cells are isolated from patients' blood and skin, cell lines are established, and genetic traits are examined.

ELIGIBILITY:
* Alpha 1-antitrypsin deficiency

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: David H. Perlmutter, Study Chair — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States